CLINICAL TRIAL: NCT05528835
Title: Effect of Prior Caesarean Delivery on ICSI Outcome
Brief Title: Caesarean Section and Intracytoplasmic Sperm Injection (ICSI) Outcome
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: 0201611
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2022-08

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 22 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Women with history of previous one Caesarean section
  Interventions: Procedure: Frozen embryo transfer
- Group B: Women with history of previous normal vaginal delivery.
  Interventions: Procedure: Frozen embryo transfer

INTERVENTIONS:
Procedure: Frozen embryo transfer — All women in both groups will receive oral estradiol valerate 8 mg/ day from the second day of the menstrual cycle. Endometrial thickness will be assessed by vaginal ultrasonography at the tenth day of treatment. When endometrial thickness reached ≥ 7 mm all subjects, in addition to estrogen, they will receive progesterone vaginal suppositories 400 mg twice daily and 100 mg of progesterone intramuscularly daily. Frozen thawed embryo transfer will be at day 6 of progesterone. Estrogen and progesterone will be continued until 9-10 weeks of gestation

SUMMARY:
Although Caesarean section (CS) is often a necessary surgical intervention, it may also be associated with an increased risk of short- and long-term sequelae. It was thought that CS may increase the risk of female subfertility or even infertility. In assisted reproductive technology (ART) cycles, the process of implantation is believed to be the most important factor in determining pregnancy outcome. In view of conflicting results on the influence of a previous CS on outcomes of ART, this study will be conducted to investigate the impact of the mode of previous delivery on ICSI outcomes.

DETAILED DESCRIPTION:
The use of CS has steadily increased worldwide and will continue increasing over the current decade where both unmet need and overuse are expected to coexist. The medical field now acknowledges a patient's right to actively participate in her choice of medical treatments, including the method of delivery what is known as CS on demand, a primary CS performed on the mother's request without any recognized medical or obstetric Indications that may also increase the rate of C.S. Although CS is often a necessary surgical intervention, it may also be associated with an increased risk of short- and long-term sequelae eg. infection, haemorrhage and increased risk of several obstetric complications in subsequent pregnancies, including mal-placentation, Caesarean scar pregnancies, morbidly adherent placentae and uterine rupture. It was thought that CS may increase the risk of female subfertility or even infertility. The possible reasons for this impact on fertility may be related to infections, adhesions formation, placental bed disruption or other non-medical factors (age, culture, education). Different mechanisms were hypothesized to explain the detrimental uterine environment associated with the presence of CS niche, that may lead to subfertility including accumulation of intrauterine fluid, altered immunobiology, increased inflammation, distorted contractility of the uterus caused by fibrosis or interruption of the myometrial layer at the site of the niche. In ART cycles, the process of implantation is believed to be the most important factor in determining pregnancy outcome, because the embryos are directly transferred into the uterine cavity and so the tubal factor can be excluded. To date, knowledge on the influence of a previous CS on outcomes of ART is limited with different conclusions in terms of live birth, miscarriage and implantation rates. In view of these conflicting results, more adequately powered studies are warranted. Therefore, this study will be conducted to investigate the impact of the mode of previous delivery on ICSI outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 20-35years.
* BMI 18- 30.
* Women with some indications for freeze all technique as patients with high risk for developing ovarian hyperstimulation syndrome (OHSS), patients with treatable tubal or uterine anomalies that were discovered during controlled ovarian hyperstimulation (COH) or in patients with elevated serum progesterone levels

Exclusion Criteria:

* Severe form of endometriosis.
* Congenital uterine anomalies.
* Scarred uterus due to previous myomectomy.
* Women diagnosed with moderate to severe degrees of intrauterine adhesions.
* Women with fibroid uteri.
* Patients with bad quality embryos.
* Untreated hydrosalpinges.
* All fresh transfer cycles will be excluded.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women complaining of secondary infertility, whether delivered vaginally or by one previous C.S, who will undergo ICSI in the IVF private centers
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 4 weeks after embryo transfer
  The ratio between the number of gestational sacs visualized by transvaginal ultrasound and the number of transferred embryos.
Clinical pregnancy | 4 weeks after embryo transfer
  Determined by the visualization of a viable embryo within the uterine cavity by ultrasound 4 weeks after embryo transfer. Clinical pregnancy rate will be calculated as the number of clinical pregnancies divided by the number of embryo transfer procedures.

SECONDARY OUTCOMES:
Biochemical pregnancy | 11 days after embryo transfer
  Positive pregnancy test 11 days after embryos transfer followed by abnormally rising or subsequently declining human chorionic gonadotropin (hCG) levels along with the absence of a visualized gestational sac on a transvaginal ultrasound. The biochemical pregnancy rate is defined as the total number of biochemical pregnancies divided by the total number of positive pregnancy tests following an embryo transfer.
Ongoing pregnancy | 18 week after embryo transfer
  Ratio between ongoing pregnancies proceeding beyond the 20th gestational weeks to the number of embryo transfer procedures
Miscarriage rate | 18 week after embryo transfer
  Calculated as the total number of pregnancies that failed to progress after visualization of an intrauterine gestational sac divided by the total number of clinically recognized intrauterine pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed AbdElmoety El Samra, phD, Principal Investigator — Alexandria University; Mohammed Salah Abd Rabbo, PhD, Study Director — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Betran AP, Ye J, Moller AB, Souza JP, Zhang J. Trends and projections of caesarean section rates: global and regional estimates. BMJ Glob Health. 2021 Jun;6(6):e005671. doi: 10.1136/bmjgh-2021-005671. PMID 34130991
- [Background] Mylonas I, Friese K. Indications for and Risks of Elective Cesarean Section. Dtsch Arztebl Int. 2015 Jul 20;112(29-30):489-95. doi: 10.3238/arztebl.2015.0489. PMID 26249251
- [Background] Duperron L. Should patients be entitled to cesarean section on demand?: Yes. Can Fam Physician. 2011 Nov;57(11):1246, 1248, 1250 passim. No abstract available. PMID 22084452
- [Background] D'Antonio F, Timor-Tritsch IE, Palacios-Jaraquemada J, Monteagudo A, Buca D, Forlani F, Minneci G, Foti F, Manzoli L, Liberati M, Acharya G, Cali G. First-trimester detection of abnormally invasive placenta in high-risk women: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2018 Feb;51(2):176-183. doi: 10.1002/uog.18840. PMID 28833750
- [Background] O'Neill SM, Kearney PM, Kenny LC, Henriksen TB, Lutomski JE, Greene RA, Khashan AS. Caesarean delivery and subsequent pregnancy interval: a systematic review and meta-analysis. BMC Pregnancy Childbirth. 2013 Aug 27;13:165. doi: 10.1186/1471-2393-13-165. PMID 23981569
- [Background] Tollanes MC, Melve KK, Irgens LM, Skjaerven R. Reduced fertility after cesarean delivery: a maternal choice. Obstet Gynecol. 2007 Dec;110(6):1256-63. doi: 10.1097/01.AOG.0000292089.18717.9f. PMID 18055718
- [Background] Vissers J, Hehenkamp W, Lambalk CB, Huirne JA. Post-Caesarean section niche-related impaired fertility: hypothetical mechanisms. Hum Reprod. 2020 Jul 1;35(7):1484-1494. doi: 10.1093/humrep/deaa094. PMID 32613231
- [Background] Brosens JJ, Gellersen B. Something new about early pregnancy: decidual biosensoring and natural embryo selection. Ultrasound Obstet Gynecol. 2010 Jul;36(1):1-5. doi: 10.1002/uog.7714. No abstract available. PMID 20582930
- [Background] Zhao J, Hao J, Xu B, Wang Y, Li Y. Impact of previous Caesarean section on reproductive outcomes after assisted reproductive technology: systematic review and meta-analyses. Reprod Biomed Online. 2021 Aug;43(2):197-204. doi: 10.1016/j.rbmo.2021.04.007. Epub 2021 Apr 22. PMID 34253450
- [Background] Wang L, Yao W, Tang X, Yao H, Wei S, Huang J, Mol BWJ, Jin L, Yue J, Wang R. Fertility outcomes of IVF/ICSI after Caesarean section: a cohort study. Reprod Biomed Online. 2020 May;40(5):719-728. doi: 10.1016/j.rbmo.2019.12.004. Epub 2019 Dec 16. PMID 32336649
- [Background] Patounakis G, Ozcan MC, Chason RJ, Norian JM, Payson M, DeCherney AH, Yauger BJ. Impact of a prior cesarean delivery on embryo transfer: a prospective study. Fertil Steril. 2016 Aug;106(2):311-6. doi: 10.1016/j.fertnstert.2016.03.045. Epub 2016 Apr 14. PMID 27087400
- [Background] Zhang N, Chen H, Xu Z, Wang B, Sun H, Hu Y. Pregnancy, Delivery, and Neonatal Outcomes of In Vitro Fertilization-Embryo Transfer in Patient with Previous Cesarean Scar. Med Sci Monit. 2016 Sep 16;22:3288-95. doi: 10.12659/msm.900581. PMID 27636504
- [Background] Ciray HN, Aksoy T, Yaramanci K, Karayaka I, Bahceci M. In vitro culture under physiologic oxygen concentration improves blastocyst yield and quality: a prospective randomized survey on sibling oocytes. Fertil Steril. 2009 Apr;91(4 Suppl):1459-61. doi: 10.1016/j.fertnstert.2008.07.1707. Epub 2008 Aug 22. PMID 18722608